CLINICAL TRIAL: NCT04884373
Title: Patient Satiety as an Indicator of Stomach Contents and Fluid Volume: an Observational Prospective Study
Brief Title: Patient Satiety as an Indicator of Stomach Contents and Fluid Volume
Status: Completed | Type: Observational
Sponsor: Imeldaziekenhuis (Other)
Responsible Party: Principal Investigator, Peter Van de Putte, Principal investigator, MD PhD, Imeldaziekenhuis
Other Study IDs: Imelda Anesth2021-001
Record Dates: First submitted 2021-03-31; First posted 2021-05-13 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Fasting; Hunger
Keywords: Ultrasonography; Gastric ultrasound
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fasted adult patients for elective surgery: * Age ≥ 18 years
  * Fasted according to national guidelines
  * Elective surgery
  * ASA physical status I-II
  * Ability to assume both supine and right lateral decubitus position.
  * Able to understand and to sign informed consent
  Interventions: Diagnostic Test: Gastric ultrasound

INTERVENTIONS:
Diagnostic Test: Gastric ultrasound — An ultrasound exam will be performed before induction of anaesthesia. GUS results from selected patients will be systematically acquired and assessed following an algorithm (Appendix Ia). The ultrasound results will be collected on a standardized form (Appendix IIa). The technique is performed in the supine and right lateral decubitus position (Appendix Ib) and only by anesthesiologists with sufficient experience with ultrasound and the technique. The patient will be asked to indicate his/her satiety on a predetermined ten-point scale.

SUMMARY:
This research proposal aims to investigate the correlation between a) the hunger feeling as measured by a ten point scale and b) total gastric fluid volumes and content as measured with gastric PoCUS in fasted, healthy subjects > 18 of age, scheduled for elective surgery.

DETAILED DESCRIPTION:
An ultrasound exam will be performed before induction of anaesthesia. GUS results from selected patients will be systematically acquired and assessed following an algorithm (Appendix Ia). The ultrasound results will be collected on a standardized form (Appendix IIa). The technique is performed in the supine and right lateral decubitus position (Appendix Ib) and only by anesthesiologists with sufficient experience with ultrasound and the technique. The patient will be asked to indicate his/her satiety on a predetermined ten-point scale. Patient data and satiety score will be collected on a standardized form (Appendix IIb). The scanning anaesthesiologist is blinded to the result of the questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* - Age ≥ 18 years
* Fasted according to national guidelines
* Elective surgery
* ASA physical status I-II
* Ability to assume both supine and right lateral decubitus position.
* Able to understand and to sign informed consent

Exclusion Criteria:

* - Previous esophagus and gastric surgery, hiatal hernia, gastric cancer.
* Pregnancy
* Failure of GUS (defined as failure to visualize the antrum)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthy adult patients scheduled for elective surgery that fit inclusion criteria
Sampling Method: Probability Sample
Enrollment: 501 (Actual)
Dates: Start 2021-06-05 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
the correlation between total gastric fluid volume in millilitres and a ten-point (0-10) satiety scale. | Before surgery
  total gastric fluid volumes are measured with gastric point-of-care ultrasound, satiety is measured with a 0 to 10 scale. Zero stands for no satiety ( very hungry, thirsty), ten stands for fully satisfied ( no hunger or thirst).

SECONDARY OUTCOMES:
the correlation between the Perlas grading scale ( 0,1,2) and a ten-point (0-10) satiety scale. | Before surgery
  the Perlas grading scale is a semi-quantitative scale where 0 stands for no fluid appreciated in the gastric antrum with gastric ultrasound in both the supine and right lateral decubitus postion (RLD), grade 1 stands for fluid appreciated in the RLD only, grade 2 stands for fluid appreciated in both the supine and RLD position. This will be correlated to the abovementioned satiety scale.
the correlation between the type of gastric content ( no content, fluid content, solid content) and a ten-point (0-10) satiety scale | before surgery
  gastric ultrasound will reveal whether the stomach is empty, contains fluid or solid content. This will be correlated to the abovementioned satiety scale.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Van de Putte, MD PhD, Principal Investigator — Imeldaziekenhuis
Locations (1):
- Imeldaziekenhuis, Bonheiden, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Van de Putte P, Herijgers A, Wallyn A, Bleeser T, Van Dijck L, Calle B, Del Jesus Sanchez Fernandez J, Dogrul F, Hendrickx E. The correlation between patient satiety sensation and total gastric fluid volume: a prospective observational study. Can J Anaesth. 2023 Aug;70(8):1307-1314. doi: 10.1007/s12630-023-02508-0. Epub 2023 Jun 23. PMID 37353726